CLINICAL TRIAL: NCT05909943
Title: Efficacy and Safety of Ruxolitinib in Neuromyelitis Optica Spectrum Disorders
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: We are doing a clinical study of Baritinib in Neuromyelitis Optica Spectrum Disorders, similar to this one, so the study was withdrawn.
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Qiang Liu, Professor of Neurology Department, Tianjin Medical University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB2022-YX-221-01
Record Dates: First submitted 2023-03-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Neuromyelitis Optica Spectrum Disorder Relapse
MeSH Terms: interventions — ruxolitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib (Experimental): Treatment with ruxolitinib will be initiated in an initial dose regimen of 5-10 mg twice daily. Two months later, the dose of ruxolitinib will be increased to 10-15 mg twice daily.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Treatment with ruxolitinib will be initiated in an initial dose regimen of 5-10 mg twice daily. Two months later, the dose of ruxolitinib will be increased to 10-15 mg twice daily.

SUMMARY:
Neuromyelitis Optica Spectrum Disorders (NMOSD) is associated with a pathological humoral immune response against the aquaporin-4(AQP-4) water channel. Rucotinib is an oral inhibitor of JAK1 and JAK2 tyrosine kinases. It may benefit some patients with NMOSD due to the important role of JAK/STAT signaling pathway in the pathogenesis of NMOSD. Clincial trials may be needed to observe its efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients ≥ 18 years old; Diagnosis of NMO or NMO spectrum disorder according to the 2015 International diagnostic criteria for neuromyelitis optic; Clinical evidence of at least 2 relapses in last 12 months or 3 relapses in the last 24 months; EDSS <= 6.0; Rituximab should be used for at least 3 months if the condition is stable; Able and willing to give written informed consent and comply with the requirements of the study protocol.

Exclusion Criteria:

Current evidence or known history of clinically significant infection (Herpes simplex virus, varicella-zoster virus, cytomegalovirus, Epstein-Barr virus, human immunodeficiency virus, Hepatitis viruses, Syphilis, etc); Participation in another interventional trial within the last 3 months; Patients taking oral immunosuppressants such as azathioprine; Tumor disease currently or within last 5 years; Pregnant, breastfeeding, or child-bearing potential during the course of the study; Clinically relevant anemia, thrombocytopenia and dysfunction of the heart, liver, kidney or bone marrow.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
time to the first protocol-defined relapse | From baseline to one year after.
  An acute attack was defined as a new neurological worsening lasting for at least 24 hours and occurring more than 30 days after the previous attack.

SECONDARY OUTCOMES:
Worsening in EDSS | Worsening from baseline in EDSS to 52 weeks
  The Expanded Disability Status Scale (EDSS) is a rating system that is frequently used for classifying and standardizing the severity and progression. EDSS ranges from 0 to 10.
Incidence of treatment-emergent adverse events [safety and tolerability] | From baseline to 52 weeks
  Adverse events related to ruxolitinib are recorded

OTHER OUTCOMES:
Counts of peripheral blood B cell subsets | From baseline to 52 weeks
  Compare peripheral blood plasma cells before and one year after initial intervention.
Number of New, and/or Enlarging T2 Hyperintense Lesions as Detected by Optic nerve,brain and spinal cord Magnetic Resonance Imaging (MRI) | From baseline to 52 weeks
  The total number of new and/or enlarging T2 lesions for all participants was calculated as the sum of the individual number of lesions at Weeks 12, 24, and 52.
Determination of serum AQP4 antibodies | From baseline to 52 weeks
  Compare serum AQP4-ab titers before and one year after initial intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China